CLINICAL TRIAL: NCT03553342
Title: Efficacy of Oral Corticosteroid Therapy in Recurrent Paralyzes After Thyroidectomy
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: THYRCOR
Record Dates: First submitted 2018-05-23; First posted 2018-06-12 (Actual); Last update posted 2021-01-29 (Actual); Status verified 2021-01

CONDITIONS: Recurrent Paralysis of Vocal Cords
MeSH Terms: conditions — Vocal Cord Paralysis | interventions — Adrenal Cortex Hormones

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Corticoids (Experimental)
  Interventions: Drug: Corticoids
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Corticoids — Patients will receive corticosteroids therapy: 1mg/kg of prednisolone daily for seven days.
  Arms: Corticoids
Other: Placebo — Patients will receive placebo for seven days.
  Arms: Placebo

SUMMARY:
Thyroidectomy is a common surgical procedure in France. Recurrent paralysis is one of the main complications. Oral corticosteroid therapy are frequently used at a dosage of 1mg/kg for seven days, in case of recurrent paralysis to obtain remobilization as early as possible.

The main objective is to evaluate the efficacy of oral corticosteroid therapy in remobilization of vocal cords at seven days in patients with unilateral recurrent paralysis after thyroidectomy.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for simple total thyroidectomy or lobo-isthmectomy
* Patients over eighteen years old
* Free subject, whitout tutorship or curatorship or subordination
* Informed consent and signed by the patient after clear and fair information about the study.

Exclusion Criteria:

* Patients operated on a total thyroidectomy with médiastino-recurrent dissection for cancer etiology
* Patients with preoperative recurrent paralysis
* Patients with hypersensitivity to prednisolone or any of the excipients.
* Patients with contraindication to use Solupred
* Patients with anti-inflammatory of acetylsalicylic acid
* Patient with evolving virosis (hepatitis, herpes, chicken pox, zoster)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Estimated)
Dates: Start 2018-09-11 (Actual); Primary Completion 2021-09-11 (Estimated); Study Completion 2022-01-11 (Estimated)

PRIMARY OUTCOMES:
Evaluate the efficacy of oral corticosteroid in remobilization of vocal cords at seven days for patients with unilateral recurrent laryngeal nerve palsy after thyroidectomy | Seven days
  evaluated by naso fibroscope inspection

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Poitiers, Poitiers, France

REFERENCES:
- [Derived] Carvajal-Alegria E, Girault N, Donatini G, Frasca D, Tonnerre D, Cosset T, Rulliere A, Lebreton JP, Dufour X, Carsuzaa F. Oral Corticosteroids in Vocal Fold Paralysis After Thyroid Surgery: A Randomized Clinical Trial. JAMA Otolaryngol Head Neck Surg. 2025 Sep 1;151(9):874-880. doi: 10.1001/jamaoto.2025.2169. PMID 40773211